CLINICAL TRIAL: NCT02969369
Title: A Multicenter Randomized Double-blind Followed by an Open-label Extension Study to Evaluate the Efficacy, Safety, and Tolerability of SEP-363856 in Subjects With Parkinson's Disease Psychosis
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of SEP-363856 in Subjects With Parkinson's Disease Psychosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-203
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2023-06-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease Psychosis
Keywords: Parkinson's Disease Psychosis
MeSH Terms: interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEP-363856 (Experimental): SEP-363856 (25, 50, or 75mg/day), once daily
  Interventions: Drug: SEP-363856
- Placebo Capsule (Placebo Comparator): Placebo once daily
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: SEP-363856 — SEP-363856 (25, 50, or 75mg/day)
  Arms: SEP-363856
Drug: Placebo capsule — Placebo once daily
  Arms: Placebo Capsule

SUMMARY:
A study to evaluate the safety and tolerability of SEP-363856 in subjects with Parkinson's Disease Psychosis. This study is accepting male and female participants 55 years of age and older who have been diagnosed with Parkinson's Disease. This study will be conducted in 24 study centers in the United States.

The study will last approximately 21 weeks.

DETAILED DESCRIPTION:
This is a multicenter, randomized, parallel-group, placebo-controlled study evaluating the efficacy, safety, and tolerability of double-blind SEP-363856 flexibly dosed at 25, 50, or 75 mg/day for 6 weeks followed by 12 weeks of open-label extension of SEP-363856 flexibly-dosed at 25, 50, or 75 mg/day in male and female subjects ≥ 55 years of age with a clinical diagnosis of PDP. The study will randomize approximately 36 subjects to 2 treatment groups in a 2:1 ratio (approximately 24 subjects to SEP-363856 and 12 to placebo). The study will consist of 4 periods: Screening/Washout Period (up to 14 days prior to Double-blind Treatment), Double-blind Treatment Period (6 weeks), Open-label SEP-363856 Treatment Period (12 weeks), and Follow-up Period (1 week after last dose) as shown in the following figure. All postBaseline clinic visits will have a window of ± 2 days relative to the date of the Baseline visit (Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Subject, caregiver, and/or legally authorized representative understands and is willing to sign informed consent to participate in the study.
* Subject must be willing and able to comply with the study procedures and visit schedules and must be able to follow verbal and written instructions.
* Subject is male or postmenopausal female ≥ 55 years of age.
* Subject meets established diagnostic criteria for Parkinson's disease of at least one year duration, consistent with the UK Brain Bank criteria
* Subject has psychotic symptoms that began after the diagnosis of PD for at least one month, occurring at least weekly in the month prior to screening (according to subject or caregiver), and severe enough to warrant treatment with antipsychotics.
* Subject has a combined score of at least 6 or an individual score of at least 4 on the neuropsychiatric inventory (NPI) Item A (delusions) and/or Item B (hallucinations). This crieterion must be met at Visit 1 and Visit 3.
* Subject has a Mini-mental status examination (MMSE) score > 21 points out of 30.
* Subject has a caregiver (spouse or family member) who will be required to attend all visits and is able to provide study information on various scales such as the NPI.
* Subject is taking antiparkinsonian drugs or deep brain stimulation, with a stable dose/dose regimen and settings for 3 months before enrolment.
* Female subject must be postmenopausal defined as being amenorrheic for greater than two years with an appropriate clinical profile.
* Male subjects with female partner(s) of childbearing potential must agree to avoid fathering a child and use acceptable methods of birth control from screening until at least 30 days after the last study drug administration.
* Subject is, in the opinion of the Investigator, medically stable based on screening medical history, PE, neurological examination, vital signs, clinical laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, thyroid panel, and serum prolactin).
* Subject has had a stable living arrangement at the time of screening.

Exclusion Criteria:

* Subject has psychosis secondary to other toxic or metabolic disorders.
* Subject has atypical Parkinson's disease, Parkinsonism secondary to medication or other neurodegenerative disorders, such as progressive supranuclear palsy or multiple system atrophy.
* Subject has dementia diagnosed concurrent with or before Parkinson's disease, motor symptoms that began less than one year before the onset of dementia or symptoms consistent with the diagnosis of lewy body dementia (LBD), or if the psychosis occurred after ablative stereotaxic surgery.
* Subject failed 2 or more antipsychotic agents given at adequate doses for at least 4 weeks within 1 year before screening.
* Subject has had a stroke or other uncontrolled serious medical or neurological illness within 6 months of baseline.
* Subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C SSRS at Screening (ie, in the past one month), or baseline (ie, since last visit).
* Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
* Subject has participated in an investigational drug study and received investigational drug within 30 days (or longer if the half-life is known to be ≥ 150 hours) prior to the screening visit, or who is currently participating in another clinical study. Subject has previously received SEP 363856.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:
* Subject has hematological (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urological, cardiovascular, hepatic, neurologic, or allergic disease that is clinically significant or unstable (except for untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has a history of cancer or significant neoplasm.
* Subject has a disorder or history of a condition or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection, or any surgical procedure) that may interfere with drug absorption, distribution, metabolism, excretion, gastrointestinal motility, or pH, or a clinically significant abnormality of the hepatic or renal system, or a history of malabsorption.
* Subject has Alcohol or Substance Abuse Disorder (DSM 5 criteria). The only exceptions are caffeine or nicotine.
* Subject has a clinically significant abnormal 12 lead ECG that may jeopardize the subject's ability to complete the study or a screening 12 lead ECG demonstrating any one of the following: heart rate > 100 beats per minute, QRS > 120 ms, QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms (males), QTcF > 470 ms (females), or PR > 220 ms.
* Subjects with known human immunodeficiency virus (HIV) seropositivity will be excluded.
* Female subject who is pregnant or lactating.
* Subject has a presence or history of a medically diagnosed, clinically significant psychiatric disorder.
* Subject is at significant risk of harming him/herself or others according to the Investigator's judgment.
* Subject has attempted suicide within 3 months prior to screening.
* Subject has a history of allergic reaction or suspected sensitivity to any substance that is contained in the formulation.
* Subject has any clinically significant abnormal laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, thyroid panel, serum prolactin, and urine drug screen(Note: abnormal findings that may be clinically significant or of questionable significance will be discussed with the Medical Monitor prior to including subject).
* Subjects with serum alanine transaminase (ALT) or aspartate transaminase (AST) levels ≥ 3 times, serum blood urea nitrogen (BUN) or creatine ≥ 1.5 X the upper limit of the reference ranges provided by the central laboratory require retesting. If on retesting, the laboratory value remains equal to or above the ULN, the subject will be excluded.
* Subjects with a random (non-fasting) blood glucose at screening ≥ 200 mg/dL (11.1 mmol/L) and HbA1c ≥ 6.5% will be excluded.
* Subject has a prolactin concentration > 100 ng/mL at screening or has a history of pituitary adenoma.
* Subject's BMI is ≥ 30 mg/kg/m2.
* Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to first dose of study drug; has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.
* Subject consumes more than 300 mg of caffeine per day (5 cups of coffee or equivalent in caffeinated beverages).
* Subject has used disallowed prescription medications or anticipates the need for any disallowed medication during their participation in this study. Subject is a staff member or the relative of a staff member.
* Subject is in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Continuation into Open-label Extension Cirteria

* Subject must have completed the 6-week double-blind treatment.
* Subject has not taken any medication other than the study drug for the purpose of controlling PDD symptoms

  . • There has been no clinically significant change in the subject's medical condition or Parkinson's disease, in the opinion of the investigator.
* Subject has not answered "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at any time during the DB treatment period.

Ages: 55 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-31 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Neuuro-Pain Medical Center, Fresno, California
  - Keck School of Medicine of USC/ University of Southern California, Los Angeles, California
  - CiTrials, Riverside, California
  - Georgetown University Hospial, Research Pharmacy Servcies, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - UHealth at Boca Raton, Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Miami, Dept. of Neurology, Miami, Florida
  - Compass Research, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - University of Florida Parkinson's Disease and Movement Disorder's Center, Tampa, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Brian Maddux, Cincinnati, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Department of Neurology, Philadelphia, Pennsylvania
  - Inland Northwest Research, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Isaacson SH, Goldstein M, Pahwa R, Singer C, Klos K, Pucci M, Zhang Y, Crandall D, Koblan KS, Navia B; Parkinson's Psychosis TAAR1 Study Group. Ulotaront, a Trace Amine-Associated Receptor 1/Serotonin 5-HT1A Agonist, in Patients With Parkinson Disease Psychosis: A Pilot Study. Neurol Clin Pract. 2023 Aug;13(4):e200175. doi: 10.1212/CPJ.0000000000200175. Epub 2023 May 25. PMID 37273942

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (QD)
- SEP-363856: SEP-363856 (25, 50, or 75 mg/day flexible dosing QD)
Period: Study
Arm/Group | Placebo | SEP-363856
Started | 14 | 25
Modified Intent-to-Treat Population | 14 | 24
Completed | 10 | 11
Not Completed | 4 | 14
Not completed — Adverse Event | 1 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5
Not completed — WITHDRAWAL BY PI DUE TO OTHER UNDERLYING ILLNESSES | 0 | 1
Period: Double-blind Period
Arm/Group | Placebo | SEP-363856
Started | 14 (Not all subjects who completed the Double Blind period, enrolled in the Open Label period.) | 25 (Not all subjects who completed the Double Blind period, enrolled in the Open Label period.)
Modified Intent-to-Treat Population | 14 | 24
Completed | 11 | 15
Not Completed | 3 | 10
Not completed — Adverse Event | 1 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — WITHDRAWAL BY PI DUE TO OTHER UNDERLYING ILLNESSES | 0 | 1
Period: Open-label SEP-363856 Period
Arm/Group | Placebo | SEP-363856
Started | 7 (Not all subjects who completed the Double Blind period, enrolled in the Open Label period.) | 9 (Not all subjects who completed the Double Blind period, enrolled in the Open Label period.)
Completed | 6 | 5
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SEP-363856 | Total
Number analyzed (Participants) | 14 | 25 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 12 | 20 | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.8 (7.12) | 70.4 (7.31) | 70.9 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 11 | 24 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White | 12 | 24 | 36
  Asian | 0 | 1 | 1
  Other | 1 | 0 | 1
Age, Customized [Count of Participants; unit: Participants]
  >=55 - <65 years | 2 | 5 | 7
  >=65 - <75 years | 7 | 12 | 19
  >=75 years | 5 | 8 | 13
Baseline Body Mass Index (BMI) (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: One participant is missing this measurement in the data.
  kg/m^2
    number analyzed (Participants) | 13 | 25 | 38
    (all) | 24.15 (5.239) | 26.08 (4.808) | 25.42 (4.975)
Baseline Body Mass Index (BMI) Category [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 1 | 1 | 2
  >=18.5 - <25.0 kg/m^2 | 7 | 8 | 15
  >=25.0 - <30.0 kg/m^2 | 3 | 14 | 17
  >=30.0 kg/m^2 | 2 | 2 | 4
  Missing | 1 | 0 | 1
Baseline Scale for Assessment of Positive Symptoms - Parkinson's Disease (SAPS-PD) Total Score [Mean (Standard Deviation); unit: Units on a scale] — The SAPS-PD consists of seven items assessing individual symptoms (four items for hallucinations and three items for delusions), a global hallucinations item and a global delusions item. Separate items are rated from 0 (absent) to 5 (severe) so that higher values represent a worse outcome. Total score is equal to the sum of the seven items plus the global hallucinations, plus the global delusions. Therefore a total possible score on the SAPS-PD ranges from 0 to 45. Population: One participant is missing this measurement in the data.
  Units on a scale
    number analyzed (Participants) | 13 | 25 | 38
    (all) | 14.7 (8.71) | 13.3 (6.00) | 13.8 (6.96)
Baseline Scale for Assessment of Positive Symptoms - Parkinson's Disease (SAPS-PD) Delusion Subscale [Mean (Standard Deviation); unit: Units on a scale] — The SAPS-PD subscale for delusions is defined as the sum of the three items for delusions and the global delusion item. Separate items are rated from 0 (absent) to 5 (severe) so that higher values represent a worse outcome, with a range of 0 to 20. Population: One participant is missing this measurement in the data.
  Units on a scale
    number analyzed (Participants) | 13 | 25 | 38
    (all) | 2.7 (3.95) | 3.0 (4.18) | 2.9 (4.05)
Baseline Scale for Assessment of Positive Symptoms - Parkinson's (SAPS-PD) Hallucination Subscale [Mean (Standard Deviation); unit: Units on a scale] — The SAPS-PD subscale for hallucinations is defined as the sum of the 4 items for hallucinations and the global hallucination item. Separate items are rated from 0 (absent) to 5 (severe) so that higher values represent a worse outcome, with a range of 0 to 25. Population: One participant is missing this measurement in the data.
  Units on a scale
    number analyzed (Participants) | 13 | 25 | 38
    (all) | 12.0 (6.60) | 10.3 (4.54) | 10.9 (5.31)

OUTCOME MEASURES:

1. Primary Outcome: Change From Double Blind (DB) Baseline in Total Scale for Assessment of Positive Symptoms - Parkinson's Disease ( SAPS-PD) Score at Week 6
Description: There are seven items assessing individual symptoms (four items for hallucinations and three items for delusions), a global hallucinations item and a global delusions item. Separate items are rated from 0 (absent) to 5 (severe), so that higher values represent a worse outcome. Total score is equal to the sum of the seven items plus the global hallucinations, plus the global delusions. Therefore a total possible score on the SAPS-PD ranges from 0 to 45.
  The primary analysis of the primary efficacy variable will use a mixed model for repeated measures (MMRM).
Time Frame: SAPS-PD assessments during DB treatment period, Baseline and Week 6
Population: The modified intention-to-treat (mITT) population is defined as all subjects who were randomized, received at least one dose of study drug, and had a baseline and at least one post-baseline total score in SAPS-PD or NPI or CGI-S during the DB treatment period.
  The mITT population is the primary population for the efficacy analyses. Subjects are analyzed according to randomized treatment group.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 13 | 23
Units on a scale | -1.4 [-5.6 to 2.8] | -2.5 [-5.8 to 0.8]

2. Secondary Outcome: Change From Double Blind (DB) Baseline in the Clinical Global Impression-Severity of Illness (CGI-S) at Week 6.
Description: The CGI-S score is a single value, clinician-rated assessment of illness severity and ranges from 1= 'Normal, not at all ill' to 7= 'Among the most extremely ill patients'. A higher score is associated with greater illness severity.
  Analysis Method: Mixed Model Repeated Measures (MMRM)
Time Frame: CGI-S assessments during DB treatment period, Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 14 | 20
Units on a scale | -0.7 [-1.5 to 0.1] | -0.4 [-1.1 to 0.3]

3. Secondary Outcome: Change From Double Blind (DB) Baseline in Neuropsychiatric Inventory (NPI) at Week 6
Description: The NPI is a 12-item behavior rating scale composed of a structured interview of the caregiver, which assesses psychiatric disturbance. For each subdomain, both the frequency (0 to 3 scale) and the severity (0 to 4 scale) of symptoms is determined. Higher scores represent a worse outcome. The subdomain score is the product of these two measures and ranges from 0 to 12. The combined NPI score is obtained by summing all 12 sub-domain scores and therefore ranges from 0 to 144.
  Analysis Method: Mixed Model Repeated Measures (MMRM)
Time Frame: NPI assessments during DB treatment period, Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 14 | 23
Units on a scale | -17.3 [-28.3 to -6.2] | -11.5 [-20.2 to -2.8]

4. Secondary Outcome: Change From Double-blind (DB) Baseline in Mini Mental State Evaluation (MMSE) at Week 6
Description: The Mini Mental State Examination (MMSE) for Cognition is a brief instrument, used to assess cognitive function, consisting of 11 tests including orientation, memory (recent and immediate), concentration, language, and praxis. Scores range from 0 to 30, with lower scores indicating greater cognitive impairment. MMSE, the total score is the sum of all 11 tests.
  Analysis Method: Mixed Model Repeated Measures (MMRM)
Time Frame: MMSE assessments during DB treatment period, Baseline and Week 6
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 14 | 23
Units on a scale | 0.3 [-0.9 to 1.4] | -0.8 [-1.7 to 0.2]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) during the 6-week DB and 12-week OL periods by actual treatment group.
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Untoward medical occurrences that occur after first administration of study drug are considered AEs.
  Results presented are for DB + OL periods combined (all study AEs). AE counts are displayed according to the actual treatment the subject was on at the time of the event.
Arm/Group | Placebo | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/14 | 2/32
Other Adverse Events (participants affected / at risk) | 12/14 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | SEP-363856 (N=32)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | SEP-363856 (N=32)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Asthenia (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 6 (9)
Balance disorder (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 6 (10)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 3 (5)
Aggression (Psychiatric disorders) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 1 (1) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3)
Confusional state (Psychiatric disorders) | 2 (2) | 5 (5)
Delusion (Psychiatric disorders) | 0 (0) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 2 (2) | 7 (8)
Hallucination, auditory (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 3 (6)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT02969369/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/69/NCT02969369/SAP_001.pdf